CLINICAL TRIAL: NCT03625258
Title: Influence of Mutations in the Pre-core Region of Heptatis B Virus (HBV) and Its Promoter on Serum VHB Viral Load in Chronically Infected Patients
Brief Title: Mutations of the Pre-core Region of Hepatite B Virus (HBV)
Acronym: HEPATITEB
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: AOL09-DR-CASTELAIN
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis B Virus
Keywords: mutations; infected patients
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatitis B virus (HBV) infection constitutes a major public health threat worldwide. A total of 92 patients with HBeAg-negative chronic hepatitis B infection were recruited at Amiens University Hospital. The diagnostic workup included a physical examination.In conclusion, the study results confirmed that the HBV DNA level is associated with liver fibrosis status and that HBV viral load is strongly correlated with BCP and PC mutations, and it demonstrated that the impaired base pairing 1858-1896 mutations at the base of the bulge in the e encapsidation signal is independently associated with high serum HBV DNA levels.

DETAILED DESCRIPTION:
The progression of liver disease in hepatitis B virus (HBV) infection is fostered by active virus replication. Mutations in the basal core promoter (BCP) and precore (PC) regions of the HBV genome are known to have an impact on viral replication. The aim of the present study was to assess the correlation of mutation profiles in the BCP and PC regions with the viral load in HBeAgnegative chronically infected patients. The HBV genotype, BCP/PC mutations, serum HBV DNA levels, and associated serological markers were analyzed in 92 HBeAgnegative chronically infected patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients included will be chronic carriers (HBsAg + for more than 6 months) of HBV, with detectable serum viral load greater than or equal to 100 IU / mL, included in the queue followed by Drs. Dominique Capron and Eric N'Guyen-Khac.

These patients will not be on anti-HBV treatment.

Exclusion Criteria:

* Patients under 18 years old
* Patients with their hepatitis B
* Patients with HBV viral load undetectable or less than 100 IU / mL.
* Immunosuppressive treatments such as corticosteroids or other
* The co-infection with the hepatitis C and / or HIV virus
* Patients with cancer

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: the study will be carried out from the blood samples following consultations Hepatogastroenterology in the clinical follow-up of patients chronically infected with HBV. Blood samples are stored in the Virology laboratory as part of legislation on the conservation of samples during Virology analyzes.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Genotype of HBV for which the HBV viral load is a function of pre-core mutations | 2-years
  The main objective of the study is toevaluate a genotype of HBV for which the HBV viral load is a function of pre-core mutations in chronically infected patients.The HBV markers (including HBsAg, HBeAg and anti- HBe) were measured with chemiluminescent microparticle immunoassays running on an Architect system.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Castelain, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No